CLINICAL TRIAL: NCT06022367
Title: An Investigation Into the Effect of the Head Raise and Head Turn Activation Techniques on Quality of Elicited Cervical Vestibular Evoked Myogenic Potentials (cVEMPs)
Brief Title: Activation Technique in cVEMPs
Acronym: ACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LHS0016
Record Dates: First submitted 2022-11-23; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-09

CONDITIONS: Activation Technique in cVEMP Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raise-Turn Sequence (Experimental): Participant performs cVEMP twice using the head raise activation technique followed by the head turn activation technique.
  Interventions: Diagnostic Test: Head Turn Activation Technique; Diagnostic Test: Head Raise Activation Technique
- Turn-Raise Sequence (Experimental): Participant performs cVEMP twice using the head turn activation technique followed by the head raise activation technique.
  Interventions: Diagnostic Test: Head Turn Activation Technique; Diagnostic Test: Head Raise Activation Technique

INTERVENTIONS:
Diagnostic Test: Head Turn Activation Technique — Participant sat upright with head turned to the side through 45 degrees. They are presented with an auditory stimulus delivered using insert earphones and their cVEMP response is recorded using skin electrodes.
Diagnostic Test: Head Raise Activation Technique — Participant assumes caloric test position (30 degrees from horizontal) with head raised. Participant is presented with an auditory stimulus delivered using insert earphones and their cVEMP response is recorded using skin electrodes.

SUMMARY:
This study will investigate two different techniques used for eliciting sternocleidomastoid (SCM) muscle contraction. Sustained contraction of the SCM muscle is necessary for accurate recording of cervical vestibular evoked myogenic potentials (cVEMPs). These responses are used clinically to assess the function of structures within the vestibular system.

The British Society of Audiology (BSA) guidelines recommend the head turn and head raise techniques as effective methods for eliciting SCM contraction. However, they do not recommend which technique to employ, leaving that to the discretion of the clinician. The purpose of this study is to determine which activation technique to recommend in the local standard operating procedure on cVEMP testing developed by the Audiology and Vestibular Function Testing service based at the Royal Liverpool University Hospital.

Healthy volunteers will be recruited to the study. The study will be conducted at the Royal Liverpool University Hospital, Liverpool, UK.

The participants will each be invited to attend one appointment in which they will undergo cVEMP testing, performed using each activation technique in turn. After testing the participants will be asked to complete a questionnaire in which they will comment on their experience of performing each technique and assign each a tolerability rating.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Male, female or non-binary, aged 18-60 years old.

Exclusion Criteria:

* Pain, sore areas, broken skin at the sites of contact with skin electrodes
* Devices, e.g. cochlear implants, which may cause electrical interference

Exclusion criteria to cVEMP procedure :

* Conductive hearing loss of middle ear origin
* Sensitivity to sounds e.g. tinnitus, hyperacusis etc.
* Cervical spine problems

Exclusion criteria to tympanometry procedure :

* Occlusion of the external auditory canal
* Otorrhoea
* Otalgia
* Excessive wax
* Within two months of ear surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
cVEMP signal quality | During single 1.5 hour appointment
  Ratio of cVEMP signal power to background noise power

SECONDARY OUTCOMES:
cVEMP signal amplitude | During single 1.5 hour appointment
  P1-N1 amplitude measured from the P1 to N1 peaks
Activation technique tolerability rating | During single 1.5 hour appointment
  Participant reported tolerability will be scored on a four-point LIKERT scale ranging from 1 (highly intolerable) to 4 (highly tolerable)
Activation technique tolerability subjective feedback | During single 1.5 hour appointment
  Participant reported concerns shared through a post-test questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, United Kingdom